CLINICAL TRIAL: NCT03492242
Title: Monitoring of Immune Checkpoint Inhibitors Adverse Drug Reactions Through the WHO Vigilyze and French Pharmaco-vigilance Database (Base Nationale de Pharmacovigilance BNPV)
Brief Title: Immune CHeckpoint Inhibitors Monitoring of Adverse Drug ReAction
Acronym: CHIMeRA
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-18-06
Record Dates: First submitted 2018-03-28; First posted 2018-04-10 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Arthritis; Cancer; Cardiac Disease; Endocrine System Diseases; Autoimmune Diseases; Ophthalmopathy; Myositis; Neuropathy
Keywords: Anti-PD-1; Anti-PD-L1; Anti-CTLA-4; Immune checkpoint inhibitors; Immune adverse drug reactions
MeSH Terms: conditions — Arthritis; Neoplasms; Heart Diseases; Endocrine System Diseases; Autoimmune Diseases; Eye Diseases; Myositis | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adverse drug reaction induced by immune checkpoint inhibitors: Case reported in the World Health Organization (WHO) and the Base Nationale de PharmacoVigilance of patient treated by ICI, with a chronology compatible with the drug toxicity
  Interventions: Drug: Immune checkpoint inhibitor

INTERVENTIONS:
Drug: Immune checkpoint inhibitor — Immune checkpoint inhibitor targeting either PD-1, PD-L1 or CTLA-4, and included in the following list (ATC classification) as a monotherapy or in combination: Ipilimumab (L01XC11), Nivolumab (L01XC17), Pembrolizumab (L01XC18), Durvalumab (L01XC28), Avelumab (L01XC31), Atezolizumab (L01XC32).

SUMMARY:
Immune checkpoint inhibitors (ICIs) might have high grade immune-related adverse events (irAEs) from rhumatologic, endocrinologic, cardiac or other system origin. This study investigates reports of drug induced irAEs with treatment including anti-PD1, Anti-PDL-1, and Anti-CTLA4 classes using the World Health Organization (WHO) database VigiBase and the french database Base Nationale de PharmacoVigilance (BNPV).

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICIs) have dramatically improved clinical outcomes in multiple cancer types and are increasingly being tested in earlier disease settings and used in combination. However, immune-related adverse events (irAEs) can occur. Here the investigators use VigiBase (http://www.vigiaccess.org/), the World Health Organization (WHO) database of individual safety case reports, and in the Base Nationale de PharmacoVigilance (BNPV) which is the french pharmacovigilance database, to identify cases of adverse drug reaction including arthiritis, auto-immune induced diseases, cardiac diseases, endocrinologic diseases, following treatment with ICIs.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database and Base Nationale de Pharmacovigilance (BNPV) of individual safety case reports to 01/05/2018
* Adverse events reported
* Patients treated with ICIs, in monotherapy or combination, included in the ATC: Ipilimumab (L01XC11), Nivolumab (L01XC17), Pembrolizumab (L01XC18), Durvalumab (L01XC28), Avelumab (L01XC31), Atezolizumab (L01XC32).

Exclusion Criteria:

• Chronology not compatible between the drug and the toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with an ICI for a cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Adverse drug reactions induced by ICIs and reported in the World Health Organization (WHO) or the Base Nationale de Pharmacovigilance (BNPV) | Case reported in the World Health Organization (WHO) or BNPV database of individual safety case reports to May 2018
  Identification and report of cases of adverse events associated with ICIs. Drugs investigated are ICIs: Ipilimumab (L01XC11), Nivolumab (L01XC17), Pembrolizumab (L01XC18), Durvalumab (L01XC28), Avelumab (L01XC31), Atezolizumab (L01XC32).

SECONDARY OUTCOMES:
Causality assessment of reported adverse drug reaction according to the WHO system | Case reported in the World Health Organization (WHO) or BNPV database of individual safety case reports to May 2018
Description of the type of adverse drug reaction depending on the category of ICIs | Case reported in the World Health Organization (WHO) or BNPV database of individual safety case reports to May 2018
Description of the other immune related adverse events concomitant to the adverse drug reaction induced by ICIs | Case reported in the World Health Organization (WHO) or BNPV database of individual safety case reports to May 2018
Description of the duration of treatment when the toxicity happens (role of cumulative dose) | Case reported in the World Health Organization (WHO) or BNPV database of individual safety case reports to May 2018
Description of the drug-drug interactions associated with adverse events | Case reported in the World Health Organization (WHO) or BNPV database of individual safety case reports to May 2018
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed | Case reported in the World Health Organization (WHO) or BNPV database of individual safety case reports to May 2018
Description of the population of patients having adverse event | Case reported in the World Health Organization (WHO) or BNPV database of individual safety case reports to May 2018

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM., Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davis EJ, Salem JE, Young A, Green JR, Ferrell PB, Ancell KK, Lebrun-Vignes B, Moslehi JJ, Johnson DB. Hematologic Complications of Immune Checkpoint Inhibitors. Oncologist. 2019 May;24(5):584-588. doi: 10.1634/theoncologist.2018-0574. Epub 2019 Feb 28. PMID 30819785
- [Background] Salem JE, Allenbach Y, Vozy A, Brechot N, Johnson DB, Moslehi JJ, Kerneis M. Abatacept for Severe Immune Checkpoint Inhibitor-Associated Myocarditis. N Engl J Med. 2019 Jun 13;380(24):2377-2379. doi: 10.1056/NEJMc1901677. No abstract available. PMID 31189043
- [Background] Johnson DB, Manouchehri A, Haugh AM, Quach HT, Balko JM, Lebrun-Vignes B, Mammen A, Moslehi JJ, Salem JE. Neurologic toxicity associated with immune checkpoint inhibitors: a pharmacovigilance study. J Immunother Cancer. 2019 May 22;7(1):134. doi: 10.1186/s40425-019-0617-x. PMID 31118078
- [Background] Johnson DB, McDonnell WJ, Gonzalez-Ericsson PI, Al-Rohil RN, Mobley BC, Salem JE, Wang DY, Sanchez V, Wang Y, Chastain CA, Barker K, Liang Y, Warren S, Beechem JM, Menzies AM, Tio M, Long GV, Cohen JV, Guidon AC, O'Hare M, Chandra S, Chowdhary A, Lebrun-Vignes B, Goldinger SM, Rushing EJ, Buchbinder EI, Mallal SA, Shi C, Xu Y, Moslehi JJ, Sanders ME, Sosman JA, Balko JM. A case report of clonal EBV-like memory CD4+ T cell activation in fatal checkpoint inhibitor-induced encephalitis. Nat Med. 2019 Aug;25(8):1243-1250. doi: 10.1038/s41591-019-0523-2. Epub 2019 Jul 22. PMID 31332390
- [Background] Bonaca MP, Olenchock BA, Salem JE, Wiviott SD, Ederhy S, Cohen A, Stewart GC, Choueiri TK, Di Carli M, Allenbach Y, Kumbhani DJ, Heinzerling L, Amiri-Kordestani L, Lyon AR, Thavendiranathan P, Padera R, Lichtman A, Liu PP, Johnson DB, Moslehi J. Myocarditis in the Setting of Cancer Therapeutics: Proposed Case Definitions for Emerging Clinical Syndromes in Cardio-Oncology. Circulation. 2019 Jul 2;140(2):80-91. doi: 10.1161/CIRCULATIONAHA.118.034497. PMID 31390169
- [Result] Arnaud L, Lebrun-Vignes B, Salem JE. Checkpoint inhibitor-associated immune arthritis. Ann Rheum Dis. 2019 Jul;78(7):e68. doi: 10.1136/annrheumdis-2018-213470. Epub 2018 May 3. No abstract available. PMID 29724725
- [Result] Wang DY, Salem JE, Cohen JV, Chandra S, Menzer C, Ye F, Zhao S, Das S, Beckermann KE, Ha L, Rathmell WK, Ancell KK, Balko JM, Bowman C, Davis EJ, Chism DD, Horn L, Long GV, Carlino MS, Lebrun-Vignes B, Eroglu Z, Hassel JC, Menzies AM, Sosman JA, Sullivan RJ, Moslehi JJ, Johnson DB. Fatal Toxic Effects Associated With Immune Checkpoint Inhibitors: A Systematic Review and Meta-analysis. JAMA Oncol. 2018 Dec 1;4(12):1721-1728. doi: 10.1001/jamaoncol.2018.3923. PMID 30242316
- [Result] Alexandre J, Moslehi JJ, Bersell KR, Funck-Brentano C, Roden DM, Salem JE. Anticancer drug-induced cardiac rhythm disorders: Current knowledge and basic underlying mechanisms. Pharmacol Ther. 2018 Sep;189:89-103. doi: 10.1016/j.pharmthera.2018.04.009. Epub 2018 Apr 24. PMID 29698683
- [Result] Wright JJ, Salem JE, Johnson DB, Lebrun-Vignes B, Stamatouli A, Thomas JW, Herold KC, Moslehi J, Powers AC. Increased Reporting of Immune Checkpoint Inhibitor-Associated Diabetes. Diabetes Care. 2018 Dec;41(12):e150-e151. doi: 10.2337/dc18-1465. Epub 2018 Oct 10. No abstract available. PMID 30305348
- [Result] Anquetil C, Salem JE, Lebrun-Vignes B, Johnson DB, Mammen AL, Stenzel W, Leonard-Louis S, Benveniste O, Moslehi JJ, Allenbach Y. Immune Checkpoint Inhibitor-Associated Myositis: Expanding the Spectrum of Cardiac Complications of the Immunotherapy Revolution. Circulation. 2018 Aug 14;138(7):743-745. doi: 10.1161/CIRCULATIONAHA.118.035898. No abstract available. PMID 30359135
- [Derived] Nguyen LS, Raia L, Lebrun-Vignes B, Salem JE. Graft Versus Host Disease Associated with Immune Checkpoint Inhibitors: A Pharmacovigilance Study and Systematic Literature Review. Front Pharmacol. 2021 Feb 5;11:619649. doi: 10.3389/fphar.2020.619649. eCollection 2020. PMID 33613286
- [Derived] Vozy A, De Martin E, Johnson DB, Lebrun-Vignes B, Moslehi JJ, Salem JE. Increased reporting of fatal hepatitis associated with immune checkpoint inhibitors. Eur J Cancer. 2019 Dec;123:112-115. doi: 10.1016/j.ejca.2019.09.022. Epub 2019 Nov 1. No abstract available. PMID 31678768